CLINICAL TRIAL: NCT06968546
Title: Randomized Controlled Study Comparing Sufentanil and Ketamine Intranasally in the Management of Severe Acute Trauma-related Pain in Children.
Brief Title: Sufentanil Versus Ketamine Intranasally in the Management of Severe Acute Trauma-related Pain in Children.
Acronym: SUF-KET-PED
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-HPNCL-03; 2025-521075-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-24; First posted 2025-05-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Traumatology; Wounds and Injury; Fractures Bone; Analgesia; Pain; Pain Management; Acute Pain
MeSH Terms: conditions — Wounds and Injuries; Fractures, Bone; Agnosia; Pain; Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal Ketamine (Active Comparator)
  Interventions: Drug: Intranasal Ketamine (IN)
- intranasal Sufentanil (Experimental)
  Interventions: Drug: Intranasal Sufentanil

INTERVENTIONS:
Drug: Intranasal Sufentanil — After randomization, the children will receive intranasal Sufentanil .
  Arms: intranasal Sufentanil
Drug: Intranasal Ketamine (IN) — After randomization, chidren will receive intranasal Ketamine
  Arms: intranasal Ketamine

SUMMARY:
Pain is one of the most common reasons for children to attend emergency departments, particularly following traumatic injuries such as fractures, sprains, or contusions. Despite advances in medical care, severe acute pain in children is still sometimes inadequately treated. One important reason is that intravenous pain medication can be technically difficult, stressful, or delayed in paediatric patients.

Intranasal drug administration, which involves spraying medication into the nose, offers a rapid and needle-free way to relieve pain and is increasingly used in paediatric emergency care. Two medications can be administered through this route: ketamine and sufentanil. Intranasal ketamine is already widely used in children for pain management. Sufentanil is a potent opioid analgesic commonly used in adults and in anaesthesia but has been much less studied in children when administered intranasally.

The aim of this study is to compare the effectiveness and safety of intranasal sufentanil and intranasal ketamine in children aged 6 to 17 years who present to the emergency department with severe traumatic limb pain. Both medications will be given in addition to standard care, including the routine use of an oxygen-nitrous oxide gas mixture (MEOPA), which is commonly used to reduce pain and anxiety in children.

Children who take part in the study will be randomly assigned to receive either intranasal sufentanil or intranasal ketamine. Pain levels will be assessed at regular time points after medication administration using age-appropriate pain scales. Sedation level and possible side effects will also be closely monitored for a short period following treatment.

The hypothesis of this study is that intranasal sufentanil will provide greater pain relief than intranasal ketamine 30 minutes after administration, without increasing the risk of adverse effects, when both are used alongside standard emergency care.

The results of this study are expected to improve knowledge about fast, effective, and non-invasive pain relief strategies for children in emergency settings and may help optimise future pain management protocols in paediatric emergency care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 17 years inclusive, under 18 years old, weighing more than 10kg, and requiring analgesia for the management of acute pain
* Presenting with pain assessed as severe using a validated pain scale (VAS > 6/10)
* Acute traumatic lime injury
* Pain caused by trauma, excluding thoracic trauma with dyspnea and abdominal pain
* Obtaining written and signe informed consent from one of the two parents or legal guardians
* Affiliation with a social security system
* Hemodynamically stable
* For post-menarche girls: negative urine pregnancy test and effective contraception, in accordance with national regulations

Exclusion Criteria:

* Patient in a state of immediate life-threatening distress
* Parents who don't understand and/or don't speak French
* Known hypersensitivity to opiods
* Allergy to one of the study treatments
* History of epilepsy or known psychiatric illness
* History of respiratory, cardiac or renal insufficiency
* Use of serotonergic antidepressants
* Any child with an ongoing respiratory condition (asthma, laryngitis)
* Thoracic trauma
* Use of opioids within the 4 hours prior to arrival in the ermergency department
* Any child with an ongoing respiratory condition (asthma, laryngitis)
* Thoracic trauma
* Use of opioids within the 4 hours prior to arrival in the ermergency department
* History of head, abdominal, or spinal trauma
* Confirmed pregnancy
* History of toxic substance use
* Facial or nasal trauma
* Whithdrawal of informed consent from the parents or legal guardian

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity from baseline to 30 minutes after intranasal administration | 30 minutes after the administration of the treatment.
  Pain intensity will be measured using a validated 100-mm Visual Analogue Scale (VAS) appropriate for children aged 6 years and older. The baseline pain score (T0) will be recorded immediately before intranasal administration of the study medication. .

SECONDARY OUTCOMES:
Time to effective analgesia | every 5 minutes for the first 30 minutes
  Time in minutes from intranasal drug administration to the first reduction of at least 20 mm on the Visual Analogue Scale (VAS). Pain is assessed every 5 minutes up to 30 minutes. Observations are censored if rescue analgesia is required.
Excessive sedation | every 5 minutes for the first 30 minutes
  Sedation assessed using the Ramsay Sedation Scale. Excessive sedation is defined as a Ramsay score greater than 3 at any time during follow-up.
Child-reported satisfaction with pain management | at 60 minutes
  Child-reported satisfaction assessed using a smiley-face scale for children under 10 years and a validated PREM questionnaire for children aged 10 years and older.

OTHER OUTCOMES:
Adverse events | every 5 minutes for the first 30 minutes then every 10 minutes until 60 minutes after the study treatment administration.
  Occurrence of adverse events during follow-up, including respiratory depression, bradycardia, hypotension, and discomfort during intranasal administration.
Parental satisfaction with pain management | at 60 minutes
  Parental satisfaction assessed at the end of follow-up using a three-option question: satisfied, not satisfied, or no opinion.
Treatment tolerance: discomfort from intranasal instillation | every 5 minutes for the first 30 minutes then every 10 minutes until 60 minutes after the study treatment administration.
  Monitoring for potential adverse events such as discomfort from intranasal instillation. For each adverse effect, the rate of patients experiencing at least one occurrence will be calculated, the severity will be graded, and the need for additional intervention will be documented.
Treatment tolerance: Bradycardia | every 5 minutes for the first 30 minutes then every 10 minutes until 60 minutes after the study treatment administration.
  Monitoring for potential adverse events such as bradycardia. For each adverse effect, the rate of patients experiencing at least one occurrence will be calculated, the severity will be graded, and the need for additional intervention will be documented.
Treatment tolerance: Desaturation | every 5 minutes for the first 30 minutes then every 10 minutes until 60 minutes after the study treatment administration.
  Monitoring for potential adverse events such as desaturation. For each adverse effect, the rate of patients experiencing at least one occurrence will be calculated, the severity will be graded, and the need for additional intervention will be documented.
Treatment tolerance: Bradypnea | every 5 minutes for the first 30 minutes then every 10 minutes until 60 minutes after the study treatment administration.
  3 - Monitoring for potential adverse events such as bradypnea. For each adverse effect, the rate of patients experiencing at least one occurrence will be calculated, the severity will be graded, and the need for additional intervention will be documented.
Treatment tolerance: sedation | every 5 minutes for the first 30 minutes then every 10 minutes until 60 minutes after the study treatment administration.
  Monitoring for potential adverse events such as sedation. For each adverse effect, the rate of patients experiencing at least one occurrence will be calculated, the severity will be graded, and the need for additional intervention will be documented.
Assessment of supplemental analgesic consumption: Before Time 0 | Time 0
  Consumption of additional analgesics will be assessed as binary parameters (yes/no).
Assessment of supplemental analgesic consumption: After Time 0 | 60 minutes
  Consumption of additional analgesics will be assessed as binary parameters (yes/no).
Assessment of supplemental analgesic consumption: Category | 60 minutes
  3 catergories will be classified:
  * Level I (e.g., paracetamol, ibuprofen)
  * Level II (e.g., profenid)
  * MEOPA (equimolar mixture of oxygen and nitrous oxide)
Assessment of supplemental analgesic consumption: Administrative reason | 60 minutes
  The reasons for administering additional analgesics (e.g., persistent pain, child's request, clinical assessment, immobilization) will be documented.
Deadline of supplemental analgesic consumption | 60 minutes
  The time to administration of additional analgesic, defined as the time in minutes between administration of the primary treatment (T0) and the first dose of additional analgesic, will be collected and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: MARCO OLLA, MD, Principal Investigator — Fondation Lenval Hôpitaux pediatrique Nice chu Lenval
Locations (1):
- Hôpital lenval, Nice, France, France

IPD SHARING:
Plan to Share IPD: No